CLINICAL TRIAL: NCT01979237
Title: Comparing FARES Method With SPASO Method for Reduction of Anterior Shoulder Dislocation: a Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201307037RINC
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Shoulder Anterior Dislocation

ARMS (1):
- SPASO method, FARES method (Experimental): Reduction method: SPASO method, FARES method
  Interventions: Procedure: SPASO method and FARES method

INTERVENTIONS:
Procedure: SPASO method and FARES method — SPASO method and FARES method as shoulder dislocation reduction methods

SUMMARY:
Shoulder anterior dislocation is a major disease entity in emergency department. There are more than 10 reduction methods that have been reported. Traditional reduction methods require sedatives, which could cause adverse effects on the patients such as respiratory suppression and allergy. There are some reduction maneuvers reported recently which do not need sedatives prior to performing reduction, including FARES method and SPASO method. So far, there are no well-designed study to compare these two methods. Besides, in clinical experience, we found that combining these two methods could even get higher successful reduction rate. This study is aimed to compare these two methods as a prospective randomized design, and furthermore, to show that combining these two methods could get higher successful reduction rate.

ELIGIBILITY:
Inclusion Criteria:

* shoulder anterior dislocation
* conscious clear
* communicable

Exclusion Criteria:

* unconscious
* non-communicable
* humeral neck fracture
* dislocation time > 24 hours
* neurovascular compromise

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Successful reduction rate | Less than 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital (NTUH), Taipei, Taiwan

REFERENCES:
- [Derived] Lee KH, Chang SH, Hung LW. FARES and Spaso method for anterior shoulder dislocation: a prospective randomized control study demonstrating the benefit of a combined approach. Sci Rep. 2025 May 30;15(1):18974. doi: 10.1038/s41598-025-04311-x. PMID 40447745